CLINICAL TRIAL: NCT00628056
Title: Mechanisms Responsible for Cardiac and Skeletal Muscle Energetic Impairment in Diabetes
Acronym: DDCM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Prof Michael Frenneaux, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RRK3159; PG/06/104/21466
Record Dates: First submitted 2008-02-24; First posted 2008-03-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2008-02

CONDITIONS: Diabetic Cardiomyopathy
Keywords: Perhexiline; diabetes; diabetic cardiomyopathy; high energy phosphate kinetics; magnetic resonance spectroscopy
MeSH Terms: conditions — Diabetic Cardiomyopathies; Diabetes Mellitus | interventions — Perhexiline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Perhexiline
- 2 (Placebo Comparator)
  Interventions: Drug: Perhexiline

INTERVENTIONS:
Drug: Perhexiline — Intervention with Perhexiline/Placebo at 100mg twice a day for 2 weeks

SUMMARY:
Diabetes increases the risk of heart failure. This is mainly due to a disease of the blood vessels supplying the heart muscle and/or high blood pressure, but abnormal metabolism may also contribute. We plan to study the mechanisms involved in this abnormal metabolism, whilst also assessing the effects of a drug called Perhexiline which improves the abnormal metabolism that is present in diabetic patients before the development of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus(WHO definition)
* HbA1C <9
* No history of chest pain
* No evidence of Coronary Artery Disease or peripheral vascular disease
* Left ventricular ejection fraction over 50%
* No evidence of respiratory disease

Exclusion Criteria:

* Patients < 16years or who cannot provide informed consent
* Evidence of significant epicardial coronary artery disease
* Evidence of peripheral vascular disease
* Abnormal liver function tests
* Clinically apparent peripheral neuropathy
* Severe chronic renal failure (creatinine >250) or diabetic nephropathy
* Concomitant use of Amiodarone, Quinidine, Haloperidol or Selective serotonin (5HT) uptake inhibitors such as Fluoxetine and Paroxetine which may inhibit the CYP2D6 enzyme
* Patients on statin therapy for primary dyslipidemia.
* Patients with recurrent hypoglycaemia
* Women of child bearing age who are not using effective contraception (or if pregnancy test positive)

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
The primary end point of the Perhexiline intervention study will be the change in cardiac PCr/ATP ratio. | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frenneaux, MD FRCP FACC, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, Westmidlands, United Kingdom